CLINICAL TRIAL: NCT05842421
Title: Imaging Methods Like Dermoscopy, Optical Coherence Tomography, in Vivo Reflectance Confocal Microscopy and 3D Total Body Photography for the Diagnosis of Non-melanoma Skin Cancer and Its Precursors
Brief Title: Imaging Methods for the Diagnosis of Non-melanoma Skin Cancer and Its Precursors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IDNMSC
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Non-melanoma Skin Cancer
Keywords: dermoscopy; 3D total body photography; optical coherence tomography; in vivo reflectance confocal microscopy; total body photography; non-invasive imaging; confocal microscopy
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: randomized, controlled, unicentric study
Masking Description: participant and investigator, who does the clinical examination and planning of surgery are not blinded, but surgeons and pathologists are blinded to the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): After clinical examination, each lesion that is suspicious for non-melanoma skin cancer and/or its precursor, is examined with dermoscopy, optical coherence tomography, in vivo reflectance confocal microscopy and each patient gets 3D total body photography. Afterwards, decision for management of each lesion is made (excision, biopsy, local treatment or no treatment). Surgeons are blinded to the groups but get the planning of surgery of the investigator. Pathologists are blinded to the groups.
  Interventions: Device: optical coherence tomography, in vivo reflectance confocal microscopy, 3D total body photography
- Control group (No Intervention): After clinical examination, each lesion that is suspicious for non-melanoma skin cancer and/or its precursor, is examined with dermoscopy as is the standard of care. Afterwards, decision for management of each lesion is made (excision, biopsy, local treatment or no treatment). Surgeons are blinded to the groups but get the planning of surgery of the investigator. Pathologists are blinded to the groups.

INTERVENTIONS:
Device: optical coherence tomography, in vivo reflectance confocal microscopy, 3D total body photography — each lesion is in addition to examination with dermoscopy examined with optical coherence tomography, in vivo reflectance confocal microscopy, each patient is photographed with 3D total body photography
  Arms: Intervention group

SUMMARY:
Prospective, unicentric study that examines if imaging devices like total body photography, dermoscopy, optical coherence tomography and in vivo reflectance confocal microscopy as an addition to clinical examination lead to a benefit for patients in the diagnosis of non-melanoma skin cancer and their precursors

DETAILED DESCRIPTION:
250 patients with lesions that are suspicious for non-melanoma skin cancer that had not yet had a biopsy, are randomized in 2 groups. The intervention group is examined with total body photography, dermoscopy, optical coherence tomography and in vivo reflectance confocal microscopy; the control group is examined with dermoscopy only. The aim of the study is to investigate whether these methods improve the early detection of non-melanoma skin cancer and their precursors. Examined are not only the differences in management of the lesions (excision, biopsy, local treatment or no treatment) and the diagnostic accuracy of the devices.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1 or more lesions suspicious for non-melanoma skin cancer that had not yet had a biopsy or diagnostic excision of the lesions

Exclusion Criteria:

* Patients with non-melanoma skin cancer that has already been examined with a punch biopsy or diagnostic excision
* Patients younger than 18 years
* Patients that are incapable of giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Management of non-melanoma skin cancer | up to 24 months
  Is management of non-melanoma skin cancer optimized after using non-invasive imaging devices like optical coherence tomography, in vivo reflectance confocal microscopy in comparison to examination with dermoscopy alone (number of primary excisions, number of biopsies, number of secondary inpatient stays due to positive biopsies, number of local treatments and lesions in which no treatment is necessary)

SECONDARY OUTCOMES:
Comparison of diagnostic accuracy in optical coherence tomography and in vivo reflectance confocal microscopy in comparison to dermoscopy alone for non-melanoma skin cancer | up to 24 months
  Comparison of diagnostic accuracy of dermoscopy and optical coherence tomography and invivo reflectance confocal microscopy (is diagnostic accuracy of optical coherence tomography better or confocal microscopy better than in dermoscopy alone?
Diagnostic accuracy of the combination of optical coherence tomography and in vivo reflectance confocal microscopy in non-melanoma skin cancer | up to 24 months
  Does the combination of the results of optical coherence tomography and in vivo reflectance confocal microscopy in each lesion lead to an even better diagnostic accuracy than each device alone?
Diagnostic accuracy of 3D total body photography | up to 24 months
  Examination of diagnostic accuracy of 3D total body photography regarding non-melanoma skin cancer in comparison to examination with dermoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Dermatologie, Carl Gustav Carus Dresden, Medizinische Fakultät Technische Universität Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the principal investigator. The data are not publicly available due to privacy or ethical restrictions.